CLINICAL TRIAL: NCT06216782
Title: Exploring the Frontiers of Neoadjuvant Therapy for Lung Cancer: a Prospective Observational Real-world Study
Status: Recruiting | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Vice-President, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: RW-LungMate
Record Dates: First submitted 2023-12-16; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer
Keywords: Neoadjuvant therapy; Lung cancer; Long-term survival
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-small cell lung cancer patients receiving neoadjuvant therapy: Patients diagnosed with non-small cell lung cancer who received neoadjuvant therapy.
  Interventions: Other: Non-intervention
- Small cell lung cancer patients receiving neoadjuvant therapy: Patients diagnosed with small cell lung cancer who received neoadjuvant therapy.
  Interventions: Other: Non-intervention

INTERVENTIONS:
Other: Non-intervention — Non-intervention

SUMMARY:
Lung cancer is a malignant tumor with the highest incidence and mortality rate of cancer patients worldwide. Traditional treatments for lung cancer include surgery, radiotherapy and chemotherapy, etc. Although the growth and spread of the tumor can be controlled to a certain extent, the cure rate for patients with progressive stage is still low and the prognosis is poor.

Neoadjuvant therapy intends to use chemotherapy, immunotherapy, and targeted therapy to reduce the size and load of the tumor before surgery, to improve the surgical resection rate and therapeutic effect.

1. Primary research objective: to explore the therapeutic efficacy of patients with different characteristics under different neoadjuvant therapeutic regimens.
2. Secondary objectives To investigate the strengths and weaknesses of different neoadjuvant regimens in real-world clinical practice, and to investigate the long-term outcomes of patients treated with different regimens.

DETAILED DESCRIPTION:
Lung cancer is a malignant tumor with the highest incidence and mortality rate of cancer patients worldwide. Traditional treatments for lung cancer include surgery, radiotherapy and chemotherapy, etc. Although the growth and spread of the tumor can be controlled to a certain extent, the cure rate for patients with progressive stage is still low and the prognosis is poor.

Neoadjuvant therapy intends to use chemotherapy, immunotherapy, and targeted therapy to reduce the size and load of the tumor before surgery, to improve the surgical resection rate and therapeutic effect. In lung cancer treatment, neoadjuvant therapy has rate and quality of life. However, a meta-analysis confirmed that although neoadjuvant chemotherapy can significantly improve survival compared to surgery alone, with an OS HR of 0.8, the improvement in 5-year survival is only 5%. Neoadjuvant radiotherapy alone, even if it can lead to pathological remission in resected specimens, does not improve resectability or overall survival. The goal of preoperative radiotherapy is to improve OS by reducing local tumor recurrence, which is the primary goal in patients with Pancoast syndrome, for example, in whom localized lung loss has an impact on quality of life. In the literature, it has been reported that in the early treatment experience of patients with Pancoast syndrome, the percentage of incompletely resected tumors was reduced by neoadjuvant radiotherapy. The MPR or pCR rate of neoadjuvant NSCLC treatment with conventional chemotherapy and radiotherapy is less than 10%, and the improvement in 5-year overall survival is only 5%, suggesting that its efficacy is very limited.

1. Primary objective The primary objective of the study is to explore the efficacy of neoadjuvant therapy in patients with different characteristics under different neoadjuvant therapy regimens.
2. Secondary objectives To investigate the strengths and weaknesses of different neoadjuvant regimens in real-world clinical practice, and to investigate the long-term outcomes of patients treated with different regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years;
2. Pathohistologically confirmed diagnosis of non-small cell lung cancer or small cell lung cancer;
3. Received neoadjuvant therapy after diagnosis;
4. Written informed consent.

Exclusion Criteria:

1. Patients enrolled in other clinical trials;
2. Patients refused enrollment in this study;
3. Patients refused follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received neoadjuvant therapy at Shanghai Pulmonary Hospital during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-12-16 (Actual); Primary Completion 2033-12-30 (Estimated); Study Completion 2033-12-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 5 years
  The time from diagnosis until progression, recurrence, or death from any cause.

SECONDARY OUTCOMES:
Surgical conversion rate and objective response rate (ORR) | 3 to 6 months
  Surgical conversion rate: the rate of the conversion from the unresectable lung cancer before treatment to resectable after inducation therapy.
  Objective response rate (ORR): the proportion of patients with a complete response or partial response to induction therapy according to Response Evaluation Criteria in Solid Tumors (RECIST).

CONTACTS AND LOCATIONS:
Overall Officials: Peng Zhang, Ph.D., Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No